CLINICAL TRIAL: NCT07105449
Title: THC Titration of High-Potency Cannabis Concentrates: A Randomized Cross-Over Trial
Brief Title: THC Titration of High-Potency Cannabis Concentrates
Acronym: THC Titration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2024-085; 1R21DA061350-01 (NIH); 195858 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2025-05-27; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: THC
Keywords: Cannabis; THC Concentrates; Self-Titration; Subjective Effects; Cognition; THC
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: This study is a double blind, randomized, cross-over human laboratory experiment evaluating the ability of participants who regularly consume cannabis to self-titrate their THC dose when vaping high-THC liquid concentrates of different potencies (30%, 60%, 90% THC).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liquid Cannabis Concentrate (30% THC) (Experimental)
  Interventions: Drug: Cannabis (30% THC Concentrate)
- Liquid Cannabis Concentrate (60% THC) (Experimental)
  Interventions: Drug: Cannabis (60% THC Concentrate)
- Liquid Cannabis Concentrate (90% THC) (Experimental)
  Interventions: Drug: Cannabis (90% THC Concentrate)

INTERVENTIONS:
Drug: Cannabis (30% THC Concentrate) — Participants will vape 30% THC concentration of liquid cannabis ad libitum.
  Arms: Liquid Cannabis Concentrate (30% THC)
Drug: Cannabis (60% THC Concentrate) — Participants will vape 60% THC concentration of liquid cannabis ad libitum.
  Arms: Liquid Cannabis Concentrate (60% THC)
Drug: Cannabis (90% THC Concentrate) — Participants will vape 90% THC concentration of liquid cannabis ad libitum.
  Arms: Liquid Cannabis Concentrate (90% THC)

SUMMARY:
High-potency cannabis use is associated with public health risks, such as cannabis use disorder, psychotic disorders, and impaired cognition. Legal markets in the US and Canada are geared towards the commercialization of high-tetrahydrocannabinol (THC) products, including concentrates as high as 90-95%. The cannabis industry has resisted regulation of higher-potency products claiming that cannabis consumers naturally self-titrate their use, but the limited evidence to date suggests that even though consumers may use less cannabis as potency rises, consuming higher potency products still leads to greater THC consumption. The investigators will use a randomized crossover trial to evaluate the ability of 36 regular cannabis consumers (18 females and 18 males) to self-titrate the THC dose when vaping concentrates to achieve the desired psychoactive effects. The investigators will also characterize and compare the subjective, cognitive, physiological, and pharmacokinetic effects between cannabis concentrates of different potencies (30%, 60%, and 90% THC). Working with US scientists, the setting of this study will be Toronto, Canada, in the context of federal legalization of cannabis, unique access to cannabis products not available in the US for research purposes, and an encouraging regulatory environment. The investigators will test commercial products that are representative of the THC ranges available in the legal market. Aim 1: To evaluate the ability of regular cannabis consumers to self-titrate their THC dose when vaping concentrates of different potencies. The investigators will compare markers of titration (biological: THC blood levels; behavioral: inhalation topography; subjective: self-reported levels of intoxication) over a range of potencies for a comprehensive characterization of titration practice. The investigators hypothesize that participants will be able to partially but not proportionally reduce THC intake with increase in THC potency. In other words, the investigators anticipate that the proportional decrease in blood THC levels will be lower than the proportional increase in THC concentrations. Aim 2: To compare the cognitive impairment, physiological effects, and addiction liability of consuming lower versus higher THC potency concentrates. The investigators hypothesize that cognitive impairment and physiological effects will be less pronounced with lower-THC concentrates in a dose-response fashion. The investigators will also explore differences in addiction liability between potencies as higher THC concentrations may result in greater dysphoric reactions. These acute effects may be related to long term harms such as accidents, CVD events, and CUD. Exploratory Aim: To explore sex differences in titration efficiency, blood THC concentrations, cognitive impairment, physiological effects, and addiction liability. The investigators propose to analyze sex differences in our primary and secondary outcomes (e.g., whether females will be able to titrate more efficiently than males). This experimental evidence will provide data on the potential acute harms related to concentrates and inform policy decisions on the need to decrease access and/or prevent their initiation and implement information and education campaigns to increase awareness on the risks of using them.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-55 years.
* Frequency of primary exposure to cannabis 1-4 occasions per week, through any route of administration, over the past three months; participants must report experience with vaping high-potency liquid concentrates with more than 3 exposures to 90% THC and willingness to use such products in the study.
* Refrain from cannabis for 48 hours and from alcohol for 12 hours before visits.
* Agree not to drive a car for 24 hours after each visit.
* Abstain from recreational drugs for at least 48 hours prior to each visit.
* Abstain from any drugs not medically required.
* Well-controlled blood pressure for participants with hypertension.

Exclusion Criteria:

* Pregnant/breastfeeding (women of childbearing potential must have a negative pregnancy test and report use of appropriate contraception).
* Evidence of cardiac arrhythmias/failure, ischaemic heart disease.
* Recent open heart/open chest surgery or cataract surgery.
* Evidence from Structured Clinical Interview for DSM-5 [SCID-5-CT] or clinical evaluation of lifetime psychotic disorder/schizophrenia or bipolar disorder; family history of a first-degree relative with a diagnosis of psychotic disorder or schizophrenia; history of psychiatric co-morbidities in the past year (major depression, anxiety disorder or suicide attempt in past year or current suicidal ideation) and current substance use disorder/dependence.
* Evidence of neurological illness (e.g., stroke, epilepsy, traumatic brain injury).
* Renal or hepatic abnormalities (self-report and blood hematology/chemistry); and
* Respiratory diseases, including asthma and physician-diagnosed lung disease.
* Taking prescribed medications that contain either THC or cannabidiol (CBD).
* Participation in another clinical or non-therapeutic study in the last three months.
* Bleeding disorders.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (blood levels of THC and metabolites) | Before vaping, 5-min after first inhalation, and at 5-, 30-, and at 60-minute intervals until 4 hours after vaping.
  Blood concentrations (ng/mL) of THC, 11-hydroxy-Δ9-tetrahydrocannabinol (OH-THC), and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol (THC-COOH) will be collected for measurement of THC and metabolites.
  Information and comparison of the PK parameters of THC and its metabolites for each product
Inhalation Topography | During a 10-minute vaping session, participants will be asked to consume cannabis ad libitum.
  Number of puffs will be measured using the eTop device.
Inhalation Topography | During a 10-minute vaping session, participants will be asked to consume cannabis ad libitum
  puff volume (cm^3) will be measured using the eTop device.
Inhalation Topography | During a 10-minute vaping session, participants will be asked to consume cannabis ad libitum.
  puff duration (milliseconds and seconds)
Inhalation Topography | During a 10-minute vaping session, participants will be asked to consume cannabis ad libitum.
  inter and inter-puff intervals (seconds and minutes) will be measured using the eTop device

SECONDARY OUTCOMES:
Visual Analog Scales (VAS) | Before vaping, 5-min after first inhalation, and at 5-, 30-, and at 60-minute intervals until 4 hours after vaping.
  A series of Visual Analog Scales (VAS) (ranging from 0 - 100) measuring subjective effects related to liking, high, good/bad effects, and rush. Minimum total score = 0, maximum total score = 2400.
  Higher/lower scores are item dependent, therefor total score is not indicative of better/worse outcome.
Profile of Mood States (POMS) | Before vaping, and 1 hour and 2 hours after vaping.
  Used to measure high/intoxication and pleasant/unpleasant cannabis effects.
Addiction Research Centre Inventory (ARCI) | 1 hour and 2 hours after vaping
  Used to assess subjective effects of cannabis.
Cognitive Task - Sustained Attention | Before vaping and 60 minutes after vaping.
  CANTAB's Rapid Visual Information Processing test asks participants to monitor a changing series of digits and to respond only when a target sequence of digits is presented.
Cognitive Task - Visuo-Spatial Working Memory | Before vaping and 60 minutes after vaping.
  CANTAB's Spatial Working Memory test examines the maintenance and manipulation of visuospatial information.
Cognitive Task - Psychomotor Speed/Accuracy | Before vaping and 60 minutes after vaping.
  CANTAB's Cognition Kit Digit Symbol Substitution (DSST) measures rapid information processing of symbols under a time limit and has been shown to be particularly sensitive to acute cannabis administration.
Physiological Effect - Heart Rate | Before vaping, 5-min after first inhalation, and at 5-, 30-, and at 60-minute intervals until 4 hours after vaping.
  Heart rate (bpm) will be measured.
Physiological Effect - Blood Pressure | Before vaping, 5-min after first inhalation, and at 5-, 30-, and at 60-minute intervals until 4 hours after vaping.
  Systolic and diastolic blood pressure (mmHg) will be measured.
Perceived Cannabis Effects Questions | 5 hours After vaping.
  A questionnaire used to assess the perceived effects of cannabis.
Pharmacogenetic Variations | 10 minutes before vaping
  Following DNA extraction, genomic DNA will be genotyped using established methods to conduct pharmacogenomics assessments. Examples of genes with known or hypothesized roles in THC metabolism and/or response include CYP2C9 and CNR1, as well as those identified in genome-wide association studies of cannabis use traits (e.g. CHRNA2).
Sex/Gender | During baseline, prior to vaping
  Traditional Masculinity-Femininity Scale (TMF)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada